CLINICAL TRIAL: NCT02336282
Title: Feasibility and Efficacy of Transcranial Direct Current Stimulation (tDCS) and Cognitive Training for Executive Dysfunction in Adult Survivors of Childhood Acute Lymphoblastic Leukemia
Brief Title: Treatment for Executive Dysfunction in Adult Survivors of Childhood Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ALLSTIM; NCI-2015-00050 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-12-18; First posted 2015-01-12 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Adult survivor of acute lymphoblastic leukemia; Executive dysfunction; Transcranial direct current stimulation; Cancer prevention and control
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Transcranial Direct Current Stimulation; Mental Status and Dementia Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tDCS on Day 1 (Active Comparator): On day one, participants will be randomized to receive the transcranial Direct Current Stimulation (tDCS) intervention. On day two, participants receive sham intervention.
  On both days 1 and 2, within two hours of completing the intervention, participants will complete cognitive assessment.
  In the second phase of the trial, participants will be evaluated over 5 weeks using a mobile tDCS device and Brain Games Stimulation twice per week. Within two hours of completing each tDCS session, participants will complete 20 minutes of cognitive training using a mobile application installed on an iPad. Cognitive assessment will be conducted pre- and post-intervention using remote assessment.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Device: Sham; Other: Cognitive Assessment; Other: Brain Games Stimulation
- tDCS on Day 2 (Active Comparator): On day one, participants will be randomized to receive sham intervention. On day two, participants receive the transcranial Direct Current Stimulation (tDCS) intervention.
  On both days 1 and 2, within two hours of completing the intervention, participants will complete cognitive assessment.
  The second phase of the trial will be conducted the same as for participants in the tDCS on Day 1 arm. Participants will be evaluated over 5 weeks using a mobile tDCS device and Brain Games Stimulation twice per week. Within two hours of completing each tDCS session, participants will complete 20 minutes of cognitive training using a mobile application installed on an iPad. Cognitive testing will be conducted pre- and post-intervention using remote assessment.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Device: Sham; Other: Cognitive Assessment; Other: Brain Games Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — transcranial Direct Current Stimulation (tDCS) involves modulation of cerebral cortex excitability by the application of weak direct current to the scalp. tDCS is a technique that applies safe, low level direct current through large pads on the scalp to stimulate the underlying brain region, with current level < 0.10 C/cm2. Direct current is transferred by a pair of saline-soaked sponges from the anode to the cathode.
  Other Names: tDCS; Transcranial Electrical Stimulation 1x1 Clinical Trials Device; Soterix Transcranial Direct Current Stimulator Clinical Trials; Soterix Medical Device 1x1-CT
Device: Sham — The sham intervention will be used in both arms with one arm receiving the sham intervention on day 1 and the other receiving the sham intervention on day 2. The sham procedure provides the same small current during ramp up to imitate the intervention, but the current is discontinued after ramp up and no intervention is provided. Direct current is transferred by a pair of saline-soaked sponges from the anode to the cathode.
  Other Names: placebo
Other: Cognitive Assessment — Three tests will be used to evaluate cognitive function: Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, and List Sorting Working Memory Test. These measures have a computerized format and are nationally standardized.
  The Gray Oral Reading Test measures reading comprehension. Participants are asked to read a set of passages and recall specific details from the stories.
  The Woodcock Johnson Understanding Directions measures listening comprehension. Participants listen to a series of complex instructions, then follow the directions by pointing to various objects in a colored picture.
  Other Names: NIH Toolbox Cognitive Battery; Gray Oral Reading Test; Woodcock Johnson Understanding Directions
Other: Brain Games Stimulation — Cognitive exercises using the Lumosity Brain Games program will be used simultaneously with the tDCS intervention. Participants will be asked to engage in training for 20 minutes a day, two days per week over 5 weeks. This program involves cognitive exercises designed to enhance executive function and processing speed.
  Other Names: Lumosity Brain Games; www.lumosity.com

SUMMARY:
A common and potentially debilitating late effect of childhood cancer treatment is neurocognitive impairment, frequently in the domain of executive dysfunction, which can limit educational attainment, employment, and quality of life. Among the survivors of childhood acute lymphoblastic leukemia (ALL) in the SJLIFE cohort, the frequency of executive function impairment has been shown as high as 58.8%, with moderate to severe impairment as high as 33.5%, and risk for impairment increased with time from diagnosis. Given the potential of pervasive impact of neurocognitive impairment on daily life, interventions directed at reducing neurocognitive dysfunction among childhood cancer survivors with long-term follow-up are needed. This study examines the potential feasibility and efficacy of a novel intervention to improve executive function.

Primary Objectives:

* To evaluate the feasibility of a home-based intervention using Transcranial Direct Current Stimulation (tDCS) and cognitive training in adult survivors of childhood ALL participating in the SJLIFE protocol at St. Jude Children's Research Hospital (SJCRH).

Secondary Objectives:

* To estimate the efficacy of a tDCS intervention paired with cognitive training.
* To explore the short-term effect of tDCS on measures of executive function among adult survivors of childhood ALL participating in the SJLIFE protocol

DETAILED DESCRIPTION:
tDCS is a form of non-invasive brain stimulation and is a potentially useful tool to enhance cognitive function. This study uses an at-home intervention of tDCS and cognitive training and examines its potential usefulness at improving executive function in ALL survivors.

Investigators will use tDCS to apply a low electrical current to the participant's scalp in the area of the brain associated with fluent and flexible thinking. The current may make that area of the brain work better for a short period of time. During this time, the participant will play computer games designed to train the brain to work more fluently flexibly. Researchers at St. Jude Children's Research Hospital want to see if pairing the electrical stimulation with the brain games at home is a feasible method to improve cognitive abilities in long-term survivors of childhood ALL.

In the first part of this study, the short-term effect of tDCS intervention will be evaluated in the clinical setting using a randomized cross-over trial. The survivors will be randomized to receive either the tDCS intervention or Sham on day 1, with the other treatment given on day 2. Neurocognitive testing will be conducted within two hours of completing stimulation each day.

In the second part of this study, the feasibility and potential efficacy of self-administration of the tDCS intervention paired with cognitive training will be evaluated over 5 weeks. Research participants will be taught to use the mobile tDCS device and will be provided one to take home. The device will be programmed by the investigators in advance to control the intensity and duration of the stimulation. The research participants will use the device twice per week as directed. Within two hours of completing each tDCS session participants will complete 20 minutes of cognitive training using a mobile app installed on an iPad. Neurocognitive testing will be conducted pre- and post- intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current St. Jude LIFE (SJLIFE) Protocol Participant
* Long term survivor of acute lymphoblastic leukemia (ALL)
* Currently ≥ 18 years of age
* Wi-Fi internet access at home
* History of executive dysfunction, documented by neurocognitive testing, and defined as having an age-adjusted standard score <20th percentile on Trail Making Test Part B, Verbal Fluency, or Digit Span Backward.
* History of self-reported executive dysfunction in daily life, defined as having a standardized score <20th percentile on BRIEF Initiate, Shift, or Working Memory domains OR having scored <20th percentile on the Childhood Cancer Survivor Study Neurocognitive Questionnaire Task Efficiency or Memory domains.
* Participant is able to speak and understand the English language.

Exclusion Criteria:

* Any survivor with full scale intelligence quotient (IQ) <80
* Currently on stimulants or other medications intended to treat cognitive impairment
* History of seizures
* No implanted medical devices or implanted metal in the head
* Currently pregnant or planning to become pregnant.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Krull, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2015 and April 2017, 53 participants were enrolled on study to complete one session of active tDCS and one session of sham tDCS. Participants must complete both to move to the At Home tDCS phase. Twenty participants were excluded due to screening failures.
Pre-assignment Details: Participants, care providers, investigator and outcomes assessor had no knowledge of group assignment.
  During campus visit, participants received tDCS and sham sessions at day1 or day2 with only order changed due to randomization. A participant was considered as a control for him/herself. For At Home tDCS phase, single arm treatment was conducted.
Groups:
- Overall Study: Participants completed tDCS set to sham, tDCS equipment set to active condition, then were to complete 10 stimulation sessions over 5 weeks using a mobile tDCS device twice per week. Within two hours of completing each tDCS session, participants were to complete 20 minutes of cognitive training using a mobile application installed on an iPad.
Period: Overall Study
Arm/Group | Overall Study
Started | 33
Completed | 28
Not Completed | 5
Not completed — Unrelated illness | 1
Not completed — Uncomfortable with technology | 1
Not completed — Lost to Follow-up | 1
Not completed — Not enough time to complete sessions | 2

BASELINE CHARACTERISTICS:
Population: Thirty one participants completed both the tDCS equipment set to sham condition and the tDCS equipment set to active condition. Two of the 33 participants who began the overall study did not complete the second day of the campus visit. Of the 31 who completed both days of the campus visit, 28 completed the at home portion.
Groups:
- Overall Study: During campus visit, following randomized design each participant completed tDCS set to sham, tDCS equipment set to active condition, during two consecutive days. Participants who completed the campus visit session and evaluation then were to complete a single arm treatment of 10 stimulation sessions over 5 weeks using a mobile tDCS device twice per week. Within two hours of completing each tDCS session, participants were to complete 20 minutes of cognitive training using a mobile application installed on an iPad.
Arm/Group | Overall Study
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of At Home tDCS Intervention
Description: This outcome measures the feasibility of remote tDCS and cognitive training. The trial will be considered feasible if at least 50% of the survivors are able to complete 5 sessions (tDCS along with cognitive stimulation) successfully out of 10.
Time Frame: 5 weeks after participant enrollment
Population: Participant enrollment for At Home Feasibility of tDCS intervention n=28 Participants Analyzed (Week 5 reported n=25)
Measure: Count of Participants; unit: Participants
Groups:
- At Home Feasibility of tDCS Intervention: All participants completed 10 stimulation sessions over 5 weeks using a mobile tDCS device twice per week. Within two hours of completing each tDCS session, participants will complete 20 minutes of cognitive training using a mobile application installed on an iPad.
Arm/Group | At Home Feasibility of tDCS Intervention
Number analyzed (Participants) | 28
Participants | 25

2. Secondary Outcome: Digit Span Forward
Description: Digit Span Forward, Longest Digits Forward: 0-9; higher score indicates more digits recalled. Higher scores are better.
Time Frame: Baseline at participant enrollment and 5 week follow-up, results of measurements from both time points were reported in the following table.
Measure: Mean (Standard Deviation); unit: raw score
Groups:
- At Home tDCS - Baseline: Pre- At Home tDCS session
- At Home tDCS - Follow-Up: Post- At Home tDCS session
Arm/Group | At Home tDCS - Baseline | At Home tDCS - Follow-Up
Number analyzed (Participants) | 25 | 25
raw score | 5.7 (1.0) | 5.7 (0.9)

3. Secondary Outcome: Neurocognitive Questionnaire: CCSS-NCQ
Description: The CCSS-NCQ is a 25 item self-report questionnaire to assess cognitive function across multiple domains in cancer survivors. Participant responses range from 1-3 for each item with higher score indicating more problems. Domain scores are created by summing the relevant item scores for each domain. Score ranges:
  * NCQ Task Efficiency: 9-27.
  * NCQ Emotional Regulation: 3-9.
  * NCQ Organization: 3-9.
  * NCQ Memory: 4-12.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- At Home tDCS - Baseline; At Home tDCS - Follow-Up: Participants completed NCQ questionnaire examiner read
Arm/Group | At Home tDCS - Baseline | At Home tDCS - Follow-Up
Number analyzed (Participants) | 25 | 25
scores on a scale
  Task Efficiency | 17.5 (3.3) | 16.2 (4.0)
  Memory | 8.1 (2.4) | 8.3 (2.0)
  Organization | 6.1 (1.7) | 5.7 (1.6)
  Emotional Regulation | 5.9 (2.6) | 4.7 (1.6)

4. Secondary Outcome: NIH Toolbox Card Sort Task
Description: The Card Sort Task measures cognitive flexibility and attention. Pictures are presented varying along two dimensions (e.g., shape and color). Participants must sort the pictures based on a given dimension. Scores range from 0-40 with higher scores indicating better function.
Time Frame: After active and sham interventions administered on day one and day two of the trial
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- On Campus Sham tDCS: tDCS equipment set to sham condition.
- On Campus tDCS: tDCS equipment set to active condition.
Arm/Group | On Campus Sham tDCS | On Campus tDCS
Number analyzed (Participants) | 31 | 31
scores on a scale | 29.2 (0.6) | 29.1 (1.4)

5. Secondary Outcome: NIH Toolbox Flanker Task
Description: The Flanker Task measures attention and inhibitory control. Participant focuses on a given stimulus while inhibiting attention to stimuli flanking it. Scores range from 0-40 with higher scores indicating better function.
Time Frame: After active and sham interventions administered on day one and day two of the trial
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | On Campus Sham tDCS | On Campus tDCS
Number analyzed (Participants) | 31 | 31
scores on a scale | 19.9 (0.4) | 20.0 (0.0)

6. Secondary Outcome: NIH Toolbox Working Memory Function
Description: The Working Memory Task measures working memory. Participant recalls and sequences different visually and orally presented stimuli. Scores range from 0-28 with higher scores indicating better working memory.
Time Frame: After active and sham interventions administered on day one and day two of the trial
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | On Campus Sham tDCS | On Campus tDCS
Number analyzed (Participants) | 31 | 31
scores on a scale | 17.0 (3.2) | 16.8 (2.9)

7. Secondary Outcome: Digit Span Backward
Description: Digit Span Backward, Longest Digits Backward: 0-8; higher score indicates more digits recalled. Higher scores are better.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | At Home tDCS - Baseline | At Home tDCS - Follow-Up
Number analyzed (Participants) | 25 | 25
raw score | 3.7 (1.0) | 4.2 (1.0)

8. Secondary Outcome: Verbal Fluency
Description: Verbal Fluency: minimum 0 with no maximum; Count of how many words were generated in 60 seconds per letter with three letters used with no top limit. Higher scores are better.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | At Home tDCS - Baseline | At Home tDCS - Follow-Up
Number analyzed (Participants) | 25 | 25
raw score | 33.1 (11.0) | 34.7 (12.0)

9. Secondary Outcome: Oral Trail Making Part A
Description: Oral Trail Making Part A: minimum 0 with no maximum amount of time in seconds to say the given letters and numbers. Higher scores are worse.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | At Home tDCS - Baseline | At Home tDCS - Follow-Up
Number analyzed (Participants) | 25 | 25
seconds | 9.4 (2.6) | 10.0 (6.7)

10. Secondary Outcome: Oral Trail Making Part B
Description: Oral Trail Making Part B: minimum 0 with no maximum amount of time in seconds to say the given letters and numbers. Higher scores are worse.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | At Home tDCS - Baseline | At Home tDCS - Follow-Up
Number analyzed (Participants) | 25 | 25
seconds | 53.1 (38.9) | 47.2 (24.0)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored before and after every tDCS session.
Description: PRISE assesses presence of side effects for several biological systems. For each organ/function system, the participant indicates the presence of a side effect, and if present, the tolerability of the side effect (tolerable or distressing). FISER and GRSEB assess side effect impact: frequency, intensity, and burden. Each domain is rated on a 7- point Likert scale.
Groups:
- At Home tDCS: Participants completed 10 stimulation sessions over 5 weeks using a mobile tDCS device twice per week. Within two hours of completing each tDCS session, participants will complete 20 minutes of cognitive training using a mobile application installed on an iPad.
Arm/Group | On Campus Sham tDCS | On Campus tDCS | At Home tDCS
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 14/33 | 10/31 | 25/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | On Campus Sham tDCS (N=33) | On Campus tDCS (N=31) | At Home tDCS (N=28)
Ringing in Ears (Ear and labyrinth disorders) | 0 | 0 | 4
Headaches (General disorders) | 5 | 1 | 11
Fatigue/Restlessness (General disorders) | 0 | 1 | 2
Vivid Dreams/Nightmares (Psychiatric disorders) | 2 | 2 | 9
Difficulty Sleeping (Psychiatric disorders) | 0 | 1 | 4
Drowsiness During the Day (Psychiatric disorders) | 0 | 1 | 3
Itching (Skin and subcutaneous tissue disorders) | 9 | 8 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02336282/Prot_SAP_000.pdf